CLINICAL TRIAL: NCT06127394
Title: Comparison of the Efficacy of Sacral Erector Spinae Plane Block (SESPB) and Pudendal Block on Postoperative Pain and Catheter-related Bladder Discomfort (CRBD) in Patients Undergoing Trans-urethral Resection of the Prostate (TUR-P).
Brief Title: Efficacy of Sacral Erector Spinae Plane Block (SESPB) on Postoperative Pain and Catheter-related Bladder Discomfort
Acronym: SESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Bilge Olgun Keles, Assistant professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/07
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pain, Postoperative
Keywords: regional block; pudendal block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- espb group (Experimental): Block will be performed with median technique at the level of sacral 2nd vertebrae.
  Interventions: Procedure: Sacral ESP Block
- pudendal group (Active Comparator): Bilateral transperineal block will be performed
  Interventions: Procedure: Pudendal Block

INTERVENTIONS:
Procedure: Sacral ESP Block — Sacral ESPB median approach, 40 ml %0,25 Bupivacaine
  Arms: espb group
Procedure: Pudendal Block — Bilateral pudendal block, 10 ml %0,25 bupivacaine
  Arms: pudendal group

SUMMARY:
The goal of this clinical trial is to evaluate the catheter related bladder discomfort in patients who will undergoing TUR-P operation. The main questions it aims to answer are:

* Is sacral ESPB effective on the pudendal nerve dermatome?
* Is sacral ESPB as useful as pudendal block on CRBD? Participants will be divided into two groups and the first group will receive sacral espb after TUR-p operation and the second group will receive pudendal block. Investigators will be present for 24 hours

  * catheter related bladder discomfort
  * post-operative pain,
  * additional analgesic needs will be questioned and the difference between the two groups will be evaluated.

DETAILED DESCRIPTION:
This is a prospective,randomised,double-blind, single-centre,study aiming to compare the effectiveness of US guided bilateral sacral ESPB and US guided bilateral pudendal block on CRBD and pain after TUR-P. 54 patients will be included in the study and divided into two groups. All patients will be standardly monitored and will receive general anaesthesia. At the end of the cases, sacral ESPB will be applied to the first group and pudendal block to the second group, and the patients and the data questioner physician will be blinded to the study.

Primary and secondary outcomes will be questioned for 24 hours and statistics will be made according to the result.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologist (ASA) Physical status 1-3

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) Physical status 4-5
* Refused to participate in the study
* Known allergy to local anaesthetic
* Where regional anaesthesia is contraindicated
* With known neurological, haematological or muscular disease
* Patients with infection or anatomical changes in the lumbo-sacral region

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males have got prostate
Enrollment: 54 (Actual)
Dates: Start 2023-11-12 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Catheter related bladder discomfort, 0:no discomfort 4:worst discomfort | baseline ,and 24 hours
  It was evaluated with a 4-point scoring system developed and first used by Agarwall et al. . No symptoms: 0, Mild: mild discomfort that can be tolerated, Moderate: discomfort is present but not accompanied by behavioural reactions, Severe: discomfort is very severe and accompanied by body movements indicating that the patient cannot bear it.

SECONDARY OUTCOMES:
Numerical Rating Scale,0 :no pain 10:worst pain | baseline, and 24 hours
  The NRS score of the patients was "0: no pain, 10: the most severe pain experienced". An NRS value of 4 and above indicates that the pain is severe and rescue analgesia is required.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Olgun Keleş, Principal Investigator — Giresun University
Locations (1):
- Giresun Research and Training Hospital, Merkez, Giresun, Turkey (Türkiye)